CLINICAL TRIAL: NCT04053153
Title: Effects of Upper Airway Muscle Training on Obstructive Sleep Apnea Severity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Stanford University (Other)
Collaborators: Asate LLC, DE (Unknown)
Responsible Party: Principal Investigator, Clete A. Kushida, Division Chief/Medical Director, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-46406
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Will not be known if participant is getting the actual device or using the placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of musical instrument (Experimental)
  Interventions: Device: Exercise equipment (a musical instrument that is based on the Medical Didgeridoo)
- Use of sham musical instrument (Sham Comparator)
  Interventions: Device: Exercise equipment (a musical instrument that is based on the Medical Didgeridoo)

INTERVENTIONS:
Device: Exercise equipment (a musical instrument that is based on the Medical Didgeridoo) — exercise equipment (a musical instrument that is based on the Medical Didgeridoo)

SUMMARY:
The purpose of this study is to evaluate the effect of Asate Silent Sleep Training on obstructive sleep apnea (OSA) severity in patients with mild to moderate OSA. The Asate Silent Sleep Training is a muscle strengthening program that uses exercise equipment (a musical instrument that is based on the didgeridoo). The equipment is connected to an application, which provides instruction on how to perform the strengthening exercises, measures the sound produced by the musical instrument, which enables the app to provide feedback on whether the individual should blow less or more and also tracks adherence to the strengthening program.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 50
* Diagnosed by a physician with mild to moderate OSA, based upon interpretation of data recorded on a take home sleep study
* Body mass index < 30 kg/m2
* Mild to moderate OSA, AHI of 5-30

Exclusion Criteria:

1. Apnea hypopnea index on overnight sleep study > 30 per hour
2. Currently practices didgeridoo
3. Consumes more than 2 alcoholic beverages per day
4. History of chronic lung disease (e.g., COPD, asthma)
5. Oral maxillofacial issue or craniofacial musculoskeletal conditions
6. Any treatment for OSA (current or past)
7. Mobile device use frequency < once per week
8. Homelessness
9. No reliable transportation to assessment sessions
10. Planned social/family/employment obligations that would limit participant from engaging in Asate Silent Sleep training during the intervention period
11. Significant upper extremity weakness/paralysis or pain limiting ability to hold the Medical Didgeridoo
12. Uncorrected low vision or blindness
13. Deafness
14. No Internet connection/Chrome browser/mobile devices with iOS and Android
15. No USB port in computer
16. Pregnancy

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 8-12 weeks
  Apnea Hypopnea Index during sleep

IPD SHARING:
Plan to Share IPD: No